CLINICAL TRIAL: NCT05405686
Title: Endometrial Gene Expression Profiles During Ovarian Stimulation With Recombinant FSH With or Without the Addition of Recombinant LH in Genuine Poor Responders
Brief Title: Effect of LH Supplementation on the Endometrial Gene Expression Profile in Poor Ovarian Responders
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: withdrawn due to practical reasons
Sponsor: CRG UZ Brussel (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Liese Boudry, Principal investigator, CRG UZ Brussel
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: LHinPOR
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Poor Response to Ovulation Induction
Keywords: IVF; LH supplementation; endometrial gene expression
MeSH Terms: interventions — Luteinizing Hormone, beta Subunit; follitropin alfa

STUDY DESIGN:
Intervention Model Description: prospective randomized open-label cross-over study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Active Comparator): In the control group, 225 IU of recombinant FSH will be administered in a fixed antagonist protocol.
  Interventions: Drug: Follitropin alfa; Diagnostic Test: Endometrial biopsy
- Study arm (Experimental): In the study group, 225 IU of recombinant FSH plus 112,5 IU of recombinant LH will be administered.
  Interventions: Drug: Lutropin alfa; Drug: Follitropin alfa; Diagnostic Test: Endometrial biopsy

INTERVENTIONS:
Drug: Lutropin alfa — addition of recombinant luteinizing hormone
  Arms: Study arm
Drug: Follitropin alfa — recombinant follicle stimulating hormone (FSH)
Diagnostic Test: Endometrial biopsy — pipelle de cornier biopsy

SUMMARY:
This is a prospective randomized open-label cross-over study. Poor responder patients will undergo two ovarian stimulation cycles. One with recombinant follicle stimulation hormone (FSH), and an other stimulation with recombinant FSH and recombinant luteinizing hormone (LH). In both groups, a freeze-all strategy will be applied and an endometrial biopsy will be taken 7 days after final oocyte maturation trigger. Endometrial gene expression analysis will be performed on both biopsies. After completion of both treatment cycles, a frozen embryo transfer of a single embryo will be performed.

DETAILED DESCRIPTION:
This is a prospective randomized open-label cross-over study, in which patients will be randomized to either start in the control group or in the study group. Participants will undergo both treatments with an interval of minimum 1 and maximum 6 months. In both treatment arms, ovarian stimulation will be started at day 2/3 of the menstrual cycle. In the control group, 225 IU of recombinant FSH will be administered in a fixed antagonist protocol. In the study group, 225 IU of recombinant FSH plus 112,5 IU of recombinant LH will be administered. Cycle monitoring will be performed through serum estradiol (E2), progesterone (P), and luteinizing hormone (LH) assessments, combined with serial ultrasound examinations. Both groups will undergo dual triggering with gonadotropin releasing hormone agonist (GnRHa) 0,2ml and human chorionic gonadotrophin (hCG) 6500IU if one or more follicles of ≥ 17 mm are observed. The oocyte retrieval (OR) will be performed between 34 and 36 hours after final oocyte maturation trigger. At each OR, follicles will be individually meas-ured, aspirated and searched for the presence of cumulus oocyte complexes (COC). Metaphase II (MII) oocytes will then be injected to standard intra-cytoplasmatic sperm injection (ICSI) procedures. In both groups, a freeze-all strategy will be applied. An endometrial biopsy (Pipelle de Cornier ®) will be taken 7 days after final oocyte maturation trigger. After completion of both treatment cycles, a frozen embryo transfer of a single embryo will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-40 years
* Undergoing IVF/ICSI
* BMI ≥ 19 and ≤ 30
* AMH <1.2 ng/mL
* Previous conventional ovarian stimulation (OS) with < 4 metaphase II (MII) oocytes
* Regular menstrual cycle (26-35 days)
* Non-smokers
* Acceptance to do 2 consecutive ovarian stimulation cycles (between 1-6 months)
* Signed informed consent

Exclusion Criteria:

* Endometriosis > rAFS grade II
* Testicular sperm extraction
* Recurrent miscarriage (>2 previous miscarriages)
* Ovarian stimulation for pre-implantation genetic testing (PGT-A/M)
* Medical/social oocyte vitrification
* In vitro maturation (IVM)
* Untreated auto-immune, endocrine or metabolic disorders
* Asherman's syndrome

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
endometrial gene expression | 7 days after finale oocyte maturation trigger
  gene expression profile of the endometrium

SECONDARY OUTCOMES:
cumulus cell gene expression | 3-6 months
endometrial histologic analysis based on Noyes' classification system | 3-6 months
progesterone level at oocyte triggering | 3-6 months
follicular fluid (FF) hormonal analysis | 3-6 months
number of preovulatory follicles | 3-6 months
number of MII oocytes | 3-6 months
number of oocytes fertilized | 3-6 months
number of good quality embryos | 3-6 months
total dose of gonadotropins administered | 3-6 months
duration of stimulation | 3-6 months
endometrial thickness at the day of endometrial biopsy | 3-6 months
implantation rate | 6-12 months
clinical pregnancy rate | 6-12 months
live birth rate | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Blockeel, Principal Investigator — UZ Brussels

IPD SHARING:
Plan to Share IPD: Undecided